CLINICAL TRIAL: NCT03377998
Title: Expression of Erythroid Differentiation Regulator 1 (Erdr1) Cytokine in the Vitiliginous Skin Lesions: a Case Control Study
Brief Title: Expression of Erythroid Differentiation Regulator 1 (Erdr1) in Vitiligo
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Maha Fathy Elmasry, principal investigator, Cairo University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: Dermatology 4
Record Dates: First submitted 2017-12-11; First posted 2017-12-19 (Actual); Last update posted 2017-12-19 (Actual); Status verified 2017-12

CONDITIONS: Erythroid Differentiation Regulator 1 (Erdr1) Cytokine

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- vitiligo patients (Experimental): lesional skin biopsy to measure ERDR1 level
  Interventions: Other: skin biopsy
- controls (Experimental): normal skin biopsy to measure ERDR1 level
  Interventions: Other: skin biopsy

INTERVENTIONS:
Other: skin biopsy — Skin biopsy for measuring tissue levels of the Erythroid differentiation regulator 1 (Erdr1) cytokine will be taken from the lesional skin of patients of vitiligo and from normal skin of healthy controls.

SUMMARY:
Expression of Erythroid differentiation regulator 1 (Erdr1) cytokine in vitiligo

ELIGIBILITY:
Inclusion Criteria:

* Patients with generalized non-segmental vitiligo.
* Both sexes.
* Age >18 years old.
* New cases or cases not receiving any medication for at least 3 months ago.

Exclusion Criteria:

* Segmental or Universal vitiligo
* Autoimmune diseases

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2018-01 (Estimated); Primary Completion 2018-07 (Estimated); Study Completion 2018-07 (Estimated)

PRIMARY OUTCOMES:
Expression of tissue levels of erythroid differentiation regulator 1 (Erdr1) cytokine in patients of vitiligo | 6 months
  Expression of tissue levels of erythroid differentiation regulator 1 (Erdr1) cytokine in patients of vitiligo and comparing its level in normal subjects

CONTACTS AND LOCATIONS:
Overall Officials: Maha Elmasry, MD, Principal Investigator — Cairo University